CLINICAL TRIAL: NCT00444574
Title: A Phase III, Randomized, Double-Blind, Multi-Center, Parallel-Group, Placebo-Controlled, Dose Optimization Study, Designed to Evaluate the Safety and Efficacy of Methylphenidate Transdermal System (MTS) vs. CONCERTA® in Pediatric Patients Aged 6-12 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of MTS Versus Concerta in Pediatric Patients (Aged 6-12 Years) With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD485-302
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylphenidate Transdermal System (Active Comparator): Methylphenidate 2.7mg, 41.3mg, 55mg, and 82.5mg patches for 7 weeks
  Interventions: Drug: Methylphenidate Transdermal System
- Placebo (Placebo Comparator): Placebp matching MTS and Concerta for 7 weeks
  Interventions: Drug: Placebo
- Concerta (Active Comparator): Methylphenidate HCL 18mg tablet 7 weeks
  Interventions: Drug: Concerta

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — The primary objective of this study was to evaluate, under controlled conditions, the safety and efficacy of MTS compared to placebo with reference to CONCERTA
  Other Names: MTS
  Arms: Methylphenidate Transdermal System
Drug: Placebo — The primary objective of this study was to evaluate, under controlled conditions, the safety and efficacy of MTS compared to placebo with reference to CONCERTA
  Other Names: Sham treatment
  Arms: Placebo
Drug: Concerta — The primary objective of this study was to evaluate, under controlled conditions, the safety and efficacy of MTS compared to placebo with reference to CONCERTA
  Other Names: Methylphenidate HCL
  Arms: Concerta

SUMMARY:
Study designed to evaluate the safety and efficacy of MTS compared to placebo with reference to CONCERTA® in pediatric subjects diagnosed with ADHD.

DETAILED DESCRIPTION:
This is a phase III, randomized, double-blind, multi-center, parallel-group, placebo-controlled, dose optimization study designed to evaluate the safety and efficacy of MTS (12.5, 18.75, 25, and 37.5 cm2) compared to placebo with reference to CONCERTA® in pediatric subjects diagnosed with attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 6-12 years
* females of Child-bearing Potential (FOCP) must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline.
* a primary diagnosis of ADHD based on a detailed psychiatric evaluation
* a total score of =>26 on the ADHD-RS-IV at the Baseline Visit
* a minimum level of intellectual functioning, as determined by an IQ (based on KBIT) score of 80 or above
* no comorbid illness that could affect safety or tolerability or in any way interfere with the subject's participation in the study.

EXCLUSION CRITERIA:

* a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis (except ODD) with significant symptoms such as Post Traumatic Stress Disorder (PTSD), psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder
* a known non-responder to psychostimulant treatment
* overweight (Body Mass Index (BMI)-for-age >90th percentile)
* a history of seizures during the last 2 years (exclusive of infantile febrile seizures), a tic disorder, a current diagnosis and/or family history of Tourette's Disorder.
* Conduct Disorder.
* Subject has taken an investigational drug within 30 days prior to Screening.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate, under controlled conditions, the safety and efficacy of SPD485 (MTS) compared to placebo with reference to CONCERTA®, as determined by the change in the clinician completed ADHD-RS-IV at each visit. | 7 weeks

SECONDARY OUTCOMES:
CTRS-R, CPRS-R, CGI, PGA scores | 7 weeks
Treatment emergent AEs, dermal evaluations, PK | 7 weeks

REFERENCES:
- [Result] Findling RL, Bukstein OG, Melmed RD, Lopez FA, Sallee FR, Arnold LE, Pratt RD. A randomized, double-blind, placebo-controlled, parallel-group study of methylphenidate transdermal system in pediatric patients with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2008 Jan;69(1):149-59. doi: 10.4088/jcp.v69n0120. PMID 18312050
- See also: (FDA Recall Information) — http://www.fda.gov/opacom/7alerts.html